CLINICAL TRIAL: NCT01057680
Title: Potential of Resistance-Exercise and Creatine Supplementation on Aging Musculoskeletal Health
Brief Title: Effectiveness of Creatine Supplementation and Exercise on Muscle and Bone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-169
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Osteoporosis; Sarcopenia
Keywords: Bone; Muscle; Strength; Kidney; Liver; Creatine
MeSH Terms: conditions — Osteoporosis; Sarcopenia | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- creatine (Experimental): This arm will involve creatine supplementation 0.1 g per kg body mass per day while participating in a resistance training program (1 hour per day, 3 days per week).
  Interventions: Dietary Supplement: creatine monohydrate
- Sugar (Placebo Comparator): This arm will involve placebo (maltodextrin) given every day while the participant does a resistance training program (1 hour per day, 3 days per week).
  Interventions: Dietary Supplement: sugar placebo

INTERVENTIONS:
Dietary Supplement: creatine monohydrate — Powder, 0.1 g per day, 12 months
  Other Names: Rivalus
  Arms: creatine
Dietary Supplement: sugar placebo — powder, 0.1 g/day, 12 months
  Arms: Sugar

SUMMARY:
As we age, we experience a reduction in muscle and bone which inevitably decreases strength and the ability to perform tasks of daily living such as gardening, carrying groceries, and climbing stairs. Health costs associated with aging muscle and bone loss are in the billions of dollars. With the projected increase in life expectancy, the incidence of muscle and bone loss will rise and further drain the healthcare system, with greater need for hospitalization, treatment, and rehabilitation. Without effective strategies to counteract aging muscle and bone loss, we may face a healthcare crisis in the future. Creatine, a compound found in red meat and seafood, increases creatine phosphate stores in muscle, providing increased energy during high-intensity exercise. Short-term (i.e. 3-4 months) resistance-exercise and supplementation with creatine, have been shown to have a favorable effect on properties of aging muscle and bone. However, the longer-term (i.e. 1 year) effects of these interventions are unknown. Therefore, the purpose of this innovative research is to determine the longer-term effects of resistance-exercise and creatine supplementation (0.1g•kg-1) in older adults. The primary dependent variables to be assessed will include muscle hypertrophy, bone mineral and bone geometry, strength, and urinary and blood indicators of liver and kidney function. This innovative, multidisciplinary research will help contribute to the successful pursuit of prolonged independent living by improving aging musculoskeletal health for older Saskatchewan adults. Saskatchewan provides a relevant setting for this research, given the higher percentage of older adults (15%), compared to the national average (12%).

We hypothesize that creatine supplementation will increase muscle mass, strength, and bone mineral density more than placebo.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 50 years of age
* males or postmenopausal females
* not currently participating in resistance training

Exclusion Criteria:

* pre-existing kidney abnormalities
* previous fragility fractures
* history of taking medications that affect bone mineral density in the past year including bisphosphonates, parathyroid hormone, calcitonin, hormone replacement therapy, or corticosteroids (i.e. within the past year)
* suffer from severe osteoarthritis
* have taken creatine supplementation within the past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Lumbar spine bone mineral density | Baseline and 12 months

SECONDARY OUTCOMES:
Proximal femur bone mineral density | Baseline and 12 months
Whole body bone mineral density | baseline and 12 months
lean tissue mass | baseline and 12 months
Muscular strength | baseline and 12 months
Muscle thickness | baseline and 12 months
Bone speed of sound | Baseline and 12 months
bone geometry | baseline and 12 months
Complete blood count | baseline, 4 months, 8 months, 12 months
Liver enzymes | baseline, 4 months, 8 months, 12 months
kidney function (creatinine clearance) | baseline, 4 months, 8 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Darren Candow, Ph.D., Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - Faculty of Kinesiology and Health Sciences, Regina, Saskatchewan
  - College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Candow DG, Chilibeck PD, Gordon JJ, Kontulainen S. Efficacy of Creatine Supplementation and Resistance Training on Area and Density of Bone and Muscle in Older Adults. Med Sci Sports Exerc. 2021 Nov 1;53(11):2388-2395. doi: 10.1249/MSS.0000000000002722. PMID 34107512